CLINICAL TRIAL: NCT03607266
Title: Effect of Preemptive Ibuprofen and Dexketoprofen on Postoperative Opioid Consumption in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effect of Preemptive Ibuprofen and Dexketoprofen in Patients Undergoing Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Celaleddin Soyalp, Assist. prof., Yuzuncu Yil University
Other Study IDs: ibupfen
Record Dates: First submitted 2018-07-19; First posted 2018-07-31 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: ibuprofen ,; Preemptive analgesia; laparoscopic cholecystectomy; preemptive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group I (Ibuprofen): Ibuprofen Group will receive 800 mg iv ibuprofen in 100 cc of isotonic solution within 30 min before the procedure
- Group D (Dexketoprofen: Dexketoprofen Group will receive 50 mg iv dexketoprofen in addition to 100 cc of isotonic solution within 30 min before the procedure
- Placebo Group: will receive 100 cc of isotonic solution within 30 min before the procedure

SUMMARY:
The primary aim of this study is to investigate the effects of preventive ibuprofen and dexketoprofen on postoperative opioid requirement in patients undergoing elective laparoscopic cholecystectomy. The secondary aim is to compare routine administration of preemptive ibuprofen and dexketoprofen in terms of intraoperative hemodynamic parameters, postoperative complications, and patient satisfaction

DETAILED DESCRIPTION:
Study Protocol, Methodology, Procedure: The study will be conducted with 90 patients aged 18-65 years with an ASA score of I and II who are planned for elective laparoscopic cholecystectomy. Patients converted to open surgery during laparoscopy and those with an ASA score of III and IV will be excluded from the study. All the patients will undergo physical examination and laboratory tests 1 day prior to the procedure. On the same day, each patient will be informed about VAS scoring system which is based on a 0-10 scale representing the severity of pain and the patients will be asked to grade their postoperative pain on this scale, where 0 indicates no pain and 10 indicates the most severe pain.

Placebo Group will receive 100 cc of isotonic solution within 30 min before the procedure. Dexketoprofen Group will receive 50 mg iv dexketoprofen in addition to 100 cc of isotonic solution within 30 min before the procedure. Ibuprofen Group will receive 800 mg iv ibuprofen in 100 cc of isotonic solution within 30 min before the procedure. Hemodynamic parameters including heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), and oxygen saturation (SpO2) will be recorded every 10 min for each patient both preoperatively and throughout the procedure. Additionally, total operative time will be recorded for each patient. The surgical procedure will be performed under general anesthesia. Anesthetic induction will be achieved with iv 2 mg/kg propofol, 2 mcg/kg fentanyl, and 0.6 mg/kg rocuronium. Anesthetic maintenance will be achieved with 8% desflurane, 40% O2, and 1 mcg/kg fentanyl. After the surgery, deep and subcutaneous infiltration of trocar insertion sites will be achieved with 4 cc of 0.5% bupivacaine. Moreover, to antagonize the effects of muscle relaxants, intravenous 0.015 mg/kg atropine and 0.04 mg/kg neostigmine will be administered. Patient-controlled analgesia (PCA) will be adjusted to a bolus dose 25 µg of fentanyl with a maximum of 6 doses/h, lockout interval of 10 min, and no basal infusion.

Postoperative Analgesia: Intravenous PCA will be adjusted to a bolus dose 25 µg of fentanyl with a maximum of 6 doses/h, lockout interval of 10 min, and no basal infusion.

Throughout laparoscopy, an intraabdominal pressure of 12-14 mmHg will be maintained. After the procedure, the patients will be transferred to the recovery room. In the recovery room, patients with a modified Aldrete score of 9 or more will be transferred to the general ward. VAS scores at postoperative 1, 2, 4, 6, 12, and 24 h will be recorded as resting VAS scores. The nurses/physicians recording the VAS scores will be blinded to the analgesic drugs and the patient groups. Patients with a VAS score of ≥4 will receive additional 50 mg tramadol in 100 cc of isotonic solution. Total procedure time will be recorded for each patient. Postoperative events occurring within the first 24 h including nausea, vomiting, mouth dryness, itching, palpitation, and headache will be recorded for each patient. At the end of the procedure, a survey will be performed to assess patient satisfaction regarding postoperative pain and other complications. To achieve this, the patients will be asked to grade their satisfaction on a 1 to 3 scale, in which 1 represents poor, 2 represents fair, and 3 represents good outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic cholecystectomy.
* Aged 18-65 years
* ASA score of I and II.

Exclusion Criteria:

Aged under 18 year Over 65 years Failure to provide a written consent Several cardiac failure, cronic renal failure, Pregnancy, A prior known allergic reaction to the drugs to be administered, Being unable to use patient-controlled analgesia (PCA) pumps, and conversion to open surgery during laparoscopy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
opioid consumption | First 24 hours total opioid consumption
  Total opioid consumption as microgram/kg will be assessed in 24 hour surgery

CONTACTS AND LOCATIONS:
Overall Officials: CELALEDDİN SOYALP, Study Chair — Yuzuncu Yil University Dursun Odabas Medical School Anesthesiology a nd Reanimation Department, Van, Turkey
Locations (1):
- Celaleddin Soyalp, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee IO, Kim SH, Kong MH, Lee MK, Kim NS, Choi YS, Lim SH. Pain after laparoscopic cholecystectomy: the effect and timing of incisional and intraperitoneal bupivacaine. Can J Anaesth. 2001 Jun;48(6):545-50. doi: 10.1007/BF03016830. PMID 11444448